CLINICAL TRIAL: NCT06539962
Title: Interstitial Lung Disease is a Risk Factor for Cardiovascular Disease; Potential Role for Systemic Biomarkers (Krebs Von Den Lungen-6 (KL-6))
Brief Title: Interstitial Lung Disease is a Risk Factor for Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant Professor of Chest Diseases, Assiut University
Other Study IDs: WGEK72024
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Lung Disease; Cardiovascular Morbidity
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Krebs von den Lungen-6 (KL-6) — Krebs von den Lungen-6 (KL-6) will be evaluated for ability to predict cardiovascular comorbidities among IPF patients

SUMMARY:
A group of Interstitial pulmonary fibrosis will be recruited from Assiut university hospital outpatient clinic.

Evaluation will be done regarding cardiovascular comorbidities (Cardiovascular comorbidities will be evaluated with thorough assessment including; history, ECG, Lipid profile and echocardiography).

Lipid profile, CRP and KL-6 level will be assessed for recruited personnel. Regression analysis will be used to identify risk factors for cardiovascular comorbidities among IPF patients.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a chronic, progressive, parenchymal disease of the lungs. ILD has been associated with various cardiovascular co-morbidities, such as coronary artery disease (CAD) and heart failure (HF). So far, little is known regarding the cardiovascular co-morbidities in patients with idiopathic pulmonary fibrosis (IPF), the most aggressive form of ILD.

Blood biomarkers have been shown to emerging evidence in patients with IPF in clinical practice. Several blood biomarkers, including lung-epithelium specific proteins, chemokines, growth factors, proteases, and other serological markers, have been studied widely in the fields of diagnosis, disease severity, and prognosis in patients with IPF. Among them, Krebs von den Lungen-6 (KL-6) is used in clinical practice and elevated level of KL-6 is known to predict mortality in patients with IPF.

It is well documented that fibrosis is closely linked to the inflammatory response. Emerging evidence suggests that cardiac fibrosis in general is primarily due to complications associated with acute and prolonged inflammation, suggesting that even low-grade, persistent inflammation is enough to promote cardiac fibrosis. The cellular and molecular events that underpin the inflammatory processes in cardiac disease are complex and poorly understood, with many tissue and disease specific mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as Interstitial pulmonary fibrosis

Exclusion Criteria:

* Patients refusing to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Demographic characteristics of patients diagnosed with interstitial pulmonary fibrosis and recruited from Assiut university hospital outpatient clinic will be recorded, including sex, age, smoking status, underlying comorbidities, addiction status.
  Chest symptoms evaluation: Cough, expectoration, hemoptysis, dyspnea, wheeze and chest pain.
  Comorbidity evaluation; including DM, hypertension, hepatic diseases, renal diseases.
  Cardiovascular comorbidities thorough assessment including; ECG, Lipid profile and echocardiography.
  chest radiograph and computed tomography (CT) chest findings will be assessed. Laboratory investigations: Lipid profile, CRP and KL-6 level according to the manufacturer's instructions
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
percentage of patients with IPF who develop cardiovascular comorbidities | 6 months
  Prevalence, clinical pattern of cardiovascular comorbidities among Interstitial pulmonary fibrosis cases

SECONDARY OUTCOMES:
accuracy of Krebs von den Lungen-6 (KL-6) to predict cardiovascular comorbidities among Interstitial pulmonary fibrosis cases | 6 months
  accuracy of Krebs von den Lungen-6 (KL-6) to predict cardiovascular comorbidities among Interstitial pulmonary fibrosis cases

CONTACTS AND LOCATIONS:
Overall Officials: Waleed MD Gamal Elddin Khaleel, Ass. Prof., Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Agrawal A, Verma I, Shah V, Agarwal A, Sikachi RR. Cardiac manifestations of idiopathic pulmonary fibrosis. Intractable Rare Dis Res. 2016 May;5(2):70-5. doi: 10.5582/irdr.2016.01023. PMID 27195188
- [Background] Nathan SD, Basavaraj A, Reichner C, Shlobin OA, Ahmad S, Kiernan J, Burton N, Barnett SD. Prevalence and impact of coronary artery disease in idiopathic pulmonary fibrosis. Respir Med. 2010 Jul;104(7):1035-41. doi: 10.1016/j.rmed.2010.02.008. Epub 2010 Mar 2. PMID 20199856
- [Background] Stainer A, Faverio P, Busnelli S, Catalano M, Della Zoppa M, Marruchella A, Pesci A, Luppi F. Molecular Biomarkers in Idiopathic Pulmonary Fibrosis: State of the Art and Future Directions. Int J Mol Sci. 2021 Jun 10;22(12):6255. doi: 10.3390/ijms22126255. PMID 34200784